CLINICAL TRIAL: NCT01462903
Title: A Phase I Study of Adoptive Immunotherapy With Autologous Tumor Infiltrating Lymphocytes in Solid Tumors
Brief Title: A Study of Adoptive Immunotherapy With Autologous Tumor Infiltrating Lymphocytes in Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jiang Li, Sun yat-sen University cancer center, biotherapy center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SenU-200902002-2
Record Dates: First submitted 2011-09-29; First posted 2011-11-01 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Nasopharyngeal Carcinoma; Hepatocellular Carcinoma; Breast Carcinoma
Keywords: TIL; NPC; hepatocellular carcinoma; immunotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Carcinoma, Hepatocellular; Breast Neoplasms | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug, T cell immunoterhapy (Experimental)
  Interventions: Biological: tumor infiltrating lymphocytes, IL-2

INTERVENTIONS:
Biological: tumor infiltrating lymphocytes, IL-2 — Biological: Infusion of Tumor Infiltrating Lymphocytes (10e9-10e10 cells) by iv in 30 Minutes. Followed by daily sc injections of 2 MIE Interleukin-2 for two weeks.
  Other Names: TIL immunotherapy for cancers

SUMMARY:
Background: T cell based adoptive immunotherapy including CTL and TIL may stimulated the immune system and stop cancer cells from growing.

Objective: Phase I clinical trial to investigate the toxicity and immune response of therapy with autologous tumor infiltrating lymphocytes as adjuvant treatment for metastatic nasopharyngeal carcinoma and hepatocellular carcinoma after primary operation, radiotherapy and chemotherapy.

Methodology: Phase I clinical trial in patients with advanced nasopharyngeal carcinoma, hepatocellular carcinoma, breast cancer and other solid cancers. The investigators isolated lymphocytes from fresh tumor tissues, activated and expanded TILs in vitro; and infused the enough number (10e9 to 10e10) of TIL back patients.

DETAILED DESCRIPTION:
Tumor infiltrating lymphocytes were isolated from tumor tissues from tumor biopsy or operation. These TILs were cultured in human IL-2 medium for 2 to 3 weeks, and reactivated by OKT3, irradiated feeder cells from the PBMCs of healthy donors and LCL set from EBV-transformed normal B cells, and expanded in human IL-2 medium for another 15 days. 10e9 to 10e10 TILs were yielded. The phenotype, function and sterile were detected before these TILs infused patients. After accepting operation or first round of routine chemotherapy and radiotherapy, the patients were treated with autologous TILs 10e9-10e10 via intravenous in 30 min, q weekX2 weeks, and followed by two weeks with daily sc low-dose interleukine-2.

Patients will be evaluated for toxicity and immune response. Peripheral blood of patients using multimer analysis and/or ELISPOT assays. Additional, we will be able to determine anti-tumor effects from immunotherapy by evaluating the clinical response of patients with stable or progressive disease at the time of TILs infusion. Lastly, we will assess additional tumor markers in patients with relapsed/refractory disease by immunohistochemical staining of tumor sections from previous diagnostic or therapeutic biopsy samples to determine the incidence of additional tumor antigen targets that may be used in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasopharyngeal carcinoma in stage IVa or Ivb and patients with metastatic hepatocellular carcinoma were planned for tumor biopsy or primary surgeon
* Age 18 to 70 years.
* Willing to sign a durable power of attorney
* Able to understand and sign the Informed Consent Document
* Life expectancy of greater than three months
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
* Serology:

  * Seronegative for HIV antibody.
  * Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
* Hematology:

  * WBC (> 3000/mm(3)).
  * Platelet count greater than 100,000/mm.
  * Hemoglobin greater than 8.0 g/dl.
* Chemistry:

  * Serum ALT/AST less or equal to 2.5 times the upper limit of normal.
  * Serum creatinine less than or equal to 1.6 mg/dl.
  * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

Exclusion Criteria:

* Previous treatment with IL-12.
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent systemic steroid therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
• the safety and tolerability of autologous tumor infiltrating lymphocytes (TIL) in combination with Interleukin-2(IL-2) in patients with nasopharyngeal carcinoma (NPC). | {Time Frame: 12 months}
  Twenty of participants with adverse events as a measure of safety and tolerability according to standard NIH criteria including fever, mucositis, dermatitis, vomiting and hematologic toxicity leucopenia, neutropenia and lymphocytoponia etc. and a Quality of Life assessment. Adverse events will be reported on the case report form. The problility of observing at least one subject experience an adverse event in a sample of 20 subjects is 0.99, if the probability of the event occurring is assumed to be 0.2. There will be 95% power to detect a change in the proportion of adverse events in the group from 0 before treatment to 0.2 after treatment.

SECONDARY OUTCOMES:
• immune efficacy and anti-tumor effects of autologous tumor infiltrating lymphocytes (TIL) in combination with Interleukin-2(IL-2) in patients with nasopharyngeal carcinoma (NPC). | [ Time Frame: 12 Months]
  Treatment response will be measured by immune response including the frequency of EBV antigen-specific T cells and ELISPOT detection for IFNg, EBV DNA concentration and tumor size. These data will be examined for normality and transformed if required.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Xin Zeng, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University, Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Weber J, Atkins M, Hwu P, Radvanyi L, Sznol M, Yee C; Immunotherapy Task Force of the NCI Investigational Drug Steering Committee. White paper on adoptive cell therapy for cancer with tumor-infiltrating lymphocytes: a report of the CTEP subcommittee on adoptive cell therapy. Clin Cancer Res. 2011 Apr 1;17(7):1664-73. doi: 10.1158/1078-0432.CCR-10-2272. Epub 2011 Feb 15. PMID 21325070
- [Background] Dudley ME, Gross CA, Langhan MM, Garcia MR, Sherry RM, Yang JC, Phan GQ, Kammula US, Hughes MS, Citrin DE, Restifo NP, Wunderlich JR, Prieto PA, Hong JJ, Langan RC, Zlott DA, Morton KE, White DE, Laurencot CM, Rosenberg SA. CD8+ enriched "young" tumor infiltrating lymphocytes can mediate regression of metastatic melanoma. Clin Cancer Res. 2010 Dec 15;16(24):6122-31. doi: 10.1158/1078-0432.CCR-10-1297. Epub 2010 Jul 28. PMID 20668005
- [Background] Besser MJ, Shapira-Frommer R, Treves AJ, Zippel D, Itzhaki O, Schallmach E, Kubi A, Shalmon B, Hardan I, Catane R, Segal E, Markel G, Apter S, Nun AB, Kuchuk I, Shimoni A, Nagler A, Schachter J. Minimally cultured or selected autologous tumor-infiltrating lymphocytes after a lympho-depleting chemotherapy regimen in metastatic melanoma patients. J Immunother. 2009 May;32(4):415-23. doi: 10.1097/CJI.0b013e31819c8bda. PMID 19342963
- [Background] Rosenberg SA, Dudley ME. Adoptive cell therapy for the treatment of patients with metastatic melanoma. Curr Opin Immunol. 2009 Apr;21(2):233-40. doi: 10.1016/j.coi.2009.03.002. Epub 2009 Mar 21. PMID 19304471